CLINICAL TRIAL: NCT06828848
Title: An Open-label, Multicentre, Single-Arm Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of VaboremⓇ (Meropenem-Vaborbactam) in Paediatric Population With Suspected or Confirmed Gram Negative Infections, Including But Not Restricted to Complicated Urinary Tract Infections
Brief Title: A Study to Assess How Vaborem® is Taking up in the Body and Tolerated in Paediatric Patients With Gram Negative Infections, Including But Not Restricted to Complicated Urinary Tract Infections
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VABOR-KIDS-01; 2024-514656-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-09

CONDITIONS: Gram Negative Infections
Keywords: pediatric; meropenem; vaborbactam; vaborem; gram negative infection; neonate
MeSH Terms: interventions — Meropenem; vaborbactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational product arm (Experimental): Single arm study. All participants enrolled will receive the investigational product.
  Interventions: Drug: Meropenem plus vaborbactam

INTERVENTIONS:
Drug: Meropenem plus vaborbactam — Meropenem plus vaborbactam fixed dose combination adjusted by body weight up to 2g/2g

SUMMARY:
The goal of this clinical trial is to assess the pharmacokinetic (PK) and safety and tolerability of Vaborem (fixed combination of meropenem and vaborbactam) in the paediatric population aged from birth to < 18 years with suspected or confirmed Gram negative infections in need of hospitalisation and intravenous (IV) antibiotic administration.

All participants will receive Vaborem IV every 8 hours to treat the suspected or confirmed Gram negative infections for 10 up to 14 days; switch to stepdown oral antibiotic is allowed after a minimum of 3 days of Vaborem. PK sample collection will occur after at least 6 doses administration.

Participant's clinical conditions will be monitored during the entire duration of the hospitalization and during scheduled visit/s after the completion of the treatment.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent before initiation of any study-related procedures.
* Male or female, from birth to < 18 years of age, inclusive.
* Require hospitalization and a minimum of 3 days of IV antibiotic treatment for suspected or confirmed Gram negative infection as per Investigator's judgement.
* Gram negative infection, according to diagnostic criteria for complicated urinary tract infection/acute pyelonephritis (cUTI/AP), complicated intra-Abdominal Infections (cIAI), Hospital-Acquired Pneumonia/Ventilator Associated Pneumonia (HAP/VAP), Blood-Stream Infection (BSI).

Main Exclusion Criteria:

* History of any moderate or significant hypersensitivity or allergic reaction to beta-lactam antibiotics or to any component of the investigational medical product.
* Gram negative infection that in the opinion of the Investigator is unlikely to respond to the study treatment.
* In treatment with immunosuppressive agents, valproic acid, or probenecid.

Ages: 0 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) for Meropenem | Day 3
Area under the concentration-time curve (AUC) for Vaborbactam | Day 3
Maximum plasma concentration (Cmax) for Meropenem | Day 3
Maximum plasma concentration (Cmax) for Vaborbactam | Day 3
Clearance (CL) of Meropenem | Day 3
Clearance (CL) of Vaborbactam | Day 3
Half-life (t1/2) of Meropenem | Day 3
Half-life (t1/2) of Vaborbactam | Day 3
Steady-state volume of distribution (Vss) of Meropenem | Day 3
Steady-state volume of distribution (Vss) of Vaborbactam | Day 3

SECONDARY OUTCOMES:
Number of patients experiencing Treatment Emergent Adverse Events (TEAE) | From baseline (day 1) to the last follow up visit (up to day 30)

CONTACTS AND LOCATIONS:
Locations (22):
- Czechia (2):
  - Fakultni nemocnice Ostrava, Ostrava
  - Faculty Hospital Kralovske Vinohrady, Paediatric Clinic, Prague
- France (5):
  - Hôpital mère-enfant - CHU de Nantes, Nantes
  - Nice University Hospital (CHU de Nice), Nice
  - Hospital Armand Trousseau Clinical Research Site, Paris
  - Hôpital Robert Debré, Paris
  - CHRU de Tours Hôpital Clocheville Clinical Research Site, Tours
- Italy (6):
  - Policlinico di Bari, Bari
  - Ospedale Sant'Orsola, Bologna
  - Giannina Gaslini Institute, Genoa
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Ospedale Pediatrico Bambino Gesù, Rome
  - Ospedale Regina Margherita, Torino
- Poland (3):
  - Insytut Centrum Zdrowia Matki Polki / Polish Mother´s Memorial Hospital Research Institute (ICZMP), Lodz
  - Uniwersyteckie Centrum Kliniczne WUM, Warsaw
  - Wojskowy Instytut Medyczny - Państwowy Instytut Badawczy, Warsaw
- Spain (6):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Dr Josep Trueta, Girona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela